CLINICAL TRIAL: NCT02144623
Title: Pretreatment With Valproate Prior to Immunotherapy Targeting Cluster of Differentiation Antigen 20 in Chronic Lymphocytic Leukemia
Acronym: PREVAIL
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version 1.2
Record Dates: First submitted 2014-05-15; First posted 2014-05-22 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2016-09

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Valproate; Cluster of differentiation antigen 20; Lymphomas; B-cell lymphomas; Translational research; Monoclonal antibodies
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma; Lymphoma, B-Cell | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Valproate (Experimental)
  Interventions: Drug: Valproate

INTERVENTIONS:
Drug: Valproate

SUMMARY:
This trial includes patients with chronic lymphocytic leukemia, the most common kind of malignant lymphoma. Monoclonal antibodies directed against cluster of differentiation antigen 20 have improved treatment results in different forms of lymphomas; however in chronic lymphocytic leukemia treatment with monoclonal antibodies is less effective, and it has been suggested that this is depending on a lower expression of the cluster of differentiation antigen 20 protein on the chronic lymphocytic leukemia cells.

Valproate, an anticonvulsant drug, has been shown to increase the cluster of differentiation antigen 20 expression, and the rationale in this study is that an increasement of cluster of differentiation antigen 20 would make treatment with monoclonal antibodies in patients with chronic lymphocytic leukemia more effective.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Histologically confirmed chronic lymphocytic leukemia
* Leucocyte count more than 20 x 10 9/L
* No other simultaneous treatment for lymphoma
* No treatment indicated for chronic lymphocytic leukemia
* WHO performance status 0-2
* HIV negativity
* Negativity for hepatitis C virus , HBsAG, anti-hepatitis B core antigen, or other active infection uncontrolled by treatment
* Agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy
* Agree not to share study medication with another person and to return all unused study drug to the investigator
* Written informed concent

Exclusion Criteria:

* Psychiatric illness or condition which could interfere with the subjects' ability to understand the requirements of the study
* Neurological or neuropsychiatric disorder, interfering with the requirements of the study
* Hearing impairment over grade 2
* Porphyria
* History of acute or chronic hepatitis
* Family history of severe drug-induced hepatitis
* Pregnancy and lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
Levels of CD20 protein and messengerRNA in response to treatment with valproate in patients with chronic lymphatic leukemia. | Blood samples to determine the level of CD20 and messengerRNA are taken day 1 and 4 at each cycle; 3 cycles are given with a cycle length of 21 days. Valproate concentration are taken day 1, 2, 3 and 4 at each cycle.

SECONDARY OUTCOMES:
Translational blood samples. | Blood tests for translational studies of the epigenetic and transcriptional regulation of the CD20 promotor are taken prestudy, day 1, 2, 3 and 4 at each cycle and 3 months post treatment.

OTHER OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability. | During treatment period (6 weeks) and 4 weeks post treatment, in total 10 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Drott, MD, PhD, Principal Investigator — Lund University Hospital
Locations (1):
- Lund University Hospital, Department of Oncology, Lund, Sweden